CLINICAL TRIAL: NCT06706765
Title: Group Telehealth Behavioral Cough Suppression Therapy Pilot Study
Brief Title: Group Telehealth Behavioral Cough Suppression Therapy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Montana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2024-36
Record Dates: First submitted 2024-08-29; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-08

CONDITIONS: Refractory Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group Telehealth Behavioral Cough Suppression Therapy (Experimental)
  Interventions: Behavioral: Behavioral Treatment

INTERVENTIONS:
Behavioral: Behavioral Treatment — Behavioral cough suppression therapy delivered in a group setting via telehealth.

SUMMARY:
The purpose of this study is to investigate the effectiveness of behavioral cough suppression therapy (BCST) in managing refractory chronic cough (RCC) within a group telehealth setting. RCC is a cough that has lasted at least 8 weeks and has not resolved with standard medical treatment. BCST is a research-based treatment provided by specialty-trained speech-language pathologists (SLPs) for patients with RCC. Although the treatment works very well for a large proportion of patients in a standard one-on-one format, there are a limited number of SLPs available to provide this treatment and patients living in rural areas do not typically have access to an SLP trained in BCST. If BCST can effectively be delivered in a group telehealth model, it would significantly improve accessibility to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Predominantly dry cough for at least 8 weeks
* Evaluated and treated by at least one physician for cough
* Obtained a chest X-ray or chest CT scan specifically related to the cough with unremarkable results
* Access to a computer or tablet that includes a camera and able to use the device independently
* Reliable internet access
* Willing to agree to maintain confidentiality of personal information (including names) related to others in the study

Exclusion Criteria:

* Under age 18
* Coughing up blood
* Current smoker of any substance
* History of smoking or 10 or more years
* Diagnosed with a chronic lung condition (e.g., COPD, emphysema, lung cancer, idiopathic pulmonary fibrosis, chronic bronchitis, asthma)? (NOTE: If a patient has been told their cough may be (or is likely) due to asthma but they have not had any formal lung testing and asthma treatments have not helped your cough, we don't consider this a formal asthma diagnosis and will not exclude them from the study.)
* Diagnosed currently or in the past with head and neck cancer (i.e., cancer of the mouth, nose, or throat).
* Complaints of swallowing difficulty
* Taking any of the following medications, which have a known side effect of cough: Benzapril (Lotensin), Captopril (Capoten), Enalapril/Enalaprilat (Vasotec oral and injectable), Fosinopril (Monopril), Lisinopril (Zestril and Prinivil), Moexipril (Univasc), Perindopril (Aceon), Quinapril (Accupril), Ramipril (Altace), and Trandolapril (Mavik)
* Prior BCST treatment with an SLP or respiratory therapist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Leicester Cough Questionnaire | Baseline, one-week post-treatment, and one-month post-treatment
  The Leicester Cough Questionnaire is a 19-item self-report questionnaire that is valid and reliable, and repeatable every two weeks. The total possible score is 21. The higher the score the better the cough-related quality of life.

SECONDARY OUTCOMES:
Patient Global Impression of Severity Scale in Chronic Cough | Baseline, every treatment session (4-6 treatment sessions, one treatment session per week), and one-month post-treatment
  The Patient Global Impression of Severity Scale in Chronic Cough involves the patient answering the question "how do you rate your overall current cough severity?" with options of "no problem, mild, moderate, or severe problem."

CONTACTS AND LOCATIONS:
Locations (1):
- University of Montana, Missoula, Montana, United States

IPD SHARING:
Plan to Share IPD: Undecided